CLINICAL TRIAL: NCT05453409
Title: A Single-center Retrospective Study of Clinical Features, Treatment Patterns, and Survival of Sarcomas
Brief Title: Study on Clinical Features, Treatment Mode and Survival of Sarcoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, Associate chief physician, Henan Cancer Hospital
Other Study IDs: ZZUSC-11
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-12

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The clinical data of all eligible patients who received chemotherapy, radiotherapy, targeted therapy, immunotherapy, interventional therapy and surgery in Henan Tumor Hospital from June 1, 2012 to May 30, 2022 were retrospectively collected.

DETAILED DESCRIPTION:
This study was a single-center retrospective clinical study, which retrospectively collected the clinical data of all eligible patients receiving chemotherapy, radiotherapy, targeted therapy, immunotherapy, interventional therapy and surgical treatment in Henan Tumor Hospital from June 1, 2012 to May 30, 2022. The efficacy, recurrence and survival of various treatments were collected.

ELIGIBILITY:
Inclusion Criteria:

No age limit, male or female. A certain subtype of sarcoma was diagnosed by pathology in our hospital. Has received at least one hospitalization in this hospital. Target lesions can be evaluated according to solid tumor efficacy evaluation criteria (RECIST; Version 1.1) Measure diameter changes.

Complete follow-up data.

Exclusion Criteria:

No clear pathology. Incomplete follow-up data.

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sarcoma patients receiving inpatient treatment in Henan Tumor Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to approximately 24months
  Progression-free survival is defined as time from enrollment to the first occurrence of progression of disease or death from any cause within 63 days of last response assessment.
Overall survival | Up to approximately 120months
  Time from pathological diagnosis to death

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided